CLINICAL TRIAL: NCT06767878
Title: Internet Delivered Therapy for Social Anxiety in Adults (PORTiSOFIE): Study Protocol for a Randomized Controlled Trial
Brief Title: Internet Delivered Therapy for Social Anxiety in Adults
Acronym: PORTiSOFIE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Lusófona (Other)
Responsible Party: Principal Investigator, Edna Martins, Principal Investigator, Grupo Lusófona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024.03961.BD
Record Dates: First submitted 2024-12-22; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Control Group; Intervention
Keywords: Social Anxiety; internet delivered CBT; Relationship satisfaction; Sexual satisfaction
MeSH Terms: conditions — Orgasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants will have access to the treatment (PORTiSOFIE). They will have a logg in for entering the platform and acess the modules, and the measures that need to be filled throughout the study.
  Interventions: Behavioral: PORTiSOFIE
- Attention Group (Other): The control group will not receive the intervention while the experimental group goes through the protocol. Instead, they will have a weekly checkup with the therapists via the platform to monitor how they are feeling. After the experimental group finishes the intervention, if the PORTiSOFIE demonstrates preliminary indicators of effectiveness, investigators will offer it to the attention group.
  Interventions: Behavioral: PORTiSOFIE

INTERVENTIONS:
Behavioral: PORTiSOFIE — This treatment is based on the Clark and Wells model of social phobia, and it is constituted by 9 modules:
  1. Introduction of the program and overview of social anxiety disorder and symptoms
  2. Negative automatic thoughts
  3. Challenging negative automatic thoughts
  4. Behavioral experiments
  5. Exposure
  6. Exposure and self-focus attention
  7. Exposure and get closer to fears
  8. Social skill training
  9. Maintenance plan

SUMMARY:
The goal of this clinical trial is to learn if an internet-delivered CBT protocol for social anxiety in adults (PORTiSOFIE) is effective in Portugal. It will also learn about the impact that PORTiSOFIE may have on relationship dimensions of these individuals. The main questions it aims to answer are:

Does PORTiSOFIE is effective? What impact PORTiSOFIE has in relationship dimensions?

Participants will:

Be assigned to experimental group and receive intervention briefly after screening is complete; Or control group and only receive intervention after the experimental group finishes.

DETAILED DESCRIPTION:
Social Anxiety Disorder (SAD) is a common condition that affects intrapersonal (e.g., distress and impairment) and interpersonal functioning (e.g., difficulties in amorous relationships). People with SAD tend to have difficulties in communicating feelings with partners and report lower levels of relationship and sexual satisfaction. Cognitive behavioral therapy (CBT) for SAD has been found to redcuce symptoms of social anxiety, but less is known about its impact on relationship functioning. Internet-based CBT (iCBT) has gained attention for its primary advantage bridging distances and saving time for the patient. In the planned study the investigators aim to translate and culturally adapt an iCBT program for social anxiety for use in Portugal (PORTiSOFIE) and measure the effects of the program on social anxiety symptoms. The project will also study the impact on relationship satisfaction and other relevant outcomes. The investigators will conduct a randomized controlled trial and divide participants in a two-arm study with parallel groups (i.e., intervention group and wait-list group). Participants will answer questionnaires to assess social anxiety symptoms and relationship outcomes at pre-treatment, posttreatment and 6-month follow up. Participants partner's will also be asked to complete questionnaires on the same periods of time, but only regarding relationship outcomes. iCBT for SAD in adults has not yet been tested in Portugal and overall there is a gap in the literature regarding the role of partners in iCBT for SAD. The study will contribute to increase accessibility to therapy (and better mental health) by promoting online evidence-based therapies. Plus, it will help to better understand how relationship components are affected and affect clinical symptoms and their progression within receiving treatment.

ELIGIBILITY:
Inclusion Criteria for participants:

* Scores on the screening questionnaires indicating at least moderate levels of social anxiety.
* Age 18 years or over
* Fluency in Portuguese
* Access to a device with internet
* Be in a monogamous amorous relationship (regardless of sexual orientation)
* Not be receiving any ongoing treatment for social anxiety (e.g., stable antidepressants).

Inclusion Criteria for partners:

* Age 18 years or over
* Fluency in Portuguese
* Access to a device with internet.

Exclusion Criteria:

* Self-reported severe psychiatric disorders such as psychosis or personality disorder.
* Planned or ongoing medical treatments (e.g., surgery) and other personal circumstances that will interfere with the treatment (e.g., planned travel abroad).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale for Adults (LSAS) | through study completion, an average of 1 year
  It has 24 items, responded in a 4-point scale. Each item is rated regarding anxiety and avoidance, and so the total score of the scale ranges between 0 and 144, with higher scores indicating higher levels of social anxiety (i.e., below 40 - no discomfort; 40-55 - Mild social discomfort; 55-65 - Moderate social phobia; 65-80 - Marked social phobia; 80-95 - Severe social phobia; Above 95 - Very severe social phobia).
Social Phobia Inventory (SPIN) | through study completion, an average of 1 year
  Is composed by three subscales: fear, avoidance, and physical discomfort. There are 17 items in total (16 in the Portuguese version), assessing the symptoms of the previous. The scale is responded on a 4-point scale, and total score is between zero and 68, with higher scores indicating higher levels of social anxiety.
Global Measure of Relationship Satisfaction (GMREL) | through study completion, an average of 1 year
  Is constituted by 5 items responded in a 7-point Likert scale. Scores range between 5 (low relationship satisfaction) and 35 (high relationship satisfaction).
Global Measure of Sexual Satisfaction (GMSEX) | through study completion, an average of 1 year
  It has 5 items responded in a 7-point Likert scale, with total scores ranging from 5 to 25, with higher values indicating greater sexual satisfaction.

SECONDARY OUTCOMES:
Revised Dyadic Adjustment Scale (RDAS) | through study completion, an average of 1 year
  3 subscales: consensus, satisfaction, cohesion. It is a 14-item measure, that asks people to rate aspects of the relationship on a 5 or 6 point scale. Total scores range between zero and 69, with higher values indicating greater adjustment.
Inclusion of Other in the Self Scale (IOS) | through study completion, an average of 1 year
  A single-item pictorial measure, that measures how close the respondent feels with another person (in this case the amorous partner).
Difficulties in Interpersonal Emotion Regulation (DIRE) | through study completion, an average of 1 year
  It has two subscales: venting and reassurance-seeking, constituted by a total of 24 items. Three hypothetic situations are presented, and for each one, the respondent must indicate how the situation is perceived on a scale from 0 (not at all distress) to 100 (extremely distressed). Then, for each of the scenarios, is asked the likelihood (i.e., 4-point Likert scale) of responding in 7 different presented ways. Higher scores indicate higher levels of difficulties in Interpersonal emotion regulation strategies.
Personal Assessment of Intimacy in Relationships (PAIR) | through study completion, an average of 1 year
  is constituted by 36 items, responded in a 5-point Likert scale (from 1 "strongly disagree" to 5 "strongly agree"), with 18 items being reversed scored, so that higher values correspond to higher levels of intimacy. For the present study, only the communication subscale with 10 items will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Lusófona, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Investigators plan to share anonymized data on request

REFERENCES:
- [Derived] Martins EM, Pascoal PM, Pereira M, Andersson G. Internet-based therapy for social anxiety in adults in Portugal (PORTiSOFIE) and its impact on sexual and relationship satisfaction: study protocol for a randomized controlled trial. Trials. 2025 Nov 6;26(1):476. doi: 10.1186/s13063-025-09103-2. PMID 41199378